CLINICAL TRIAL: NCT04664777
Title: Intraoperative Correlation of Non Invasive Hemoglobin (SpHb) Measurement With Laboratory Hemoglobin Measurement in Living Liver Donors
Brief Title: Correlation of Non Invasive Hemoglobin Measurement With Laboratory Hemoglobin Measurement in Living Liver Donors
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yusuf Ziya ÇOLAK, Asst. Prof. Yusuf Ziya Çolak, Inonu University
Other Study IDs: Inonu universitesi
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
Keywords: hemoglobin level; Pulse CO-Oximetry; intraoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Group1: Living liver donors who operated between 1 August and 15 november:
  After anesthesia induction and surgical field sterilization, before surgical incision; blood sample will be taken, SpHb, PI and vital measurements (SpO2, Heart rate, NIBP, body temperature) will be recorded.
  After the surgical procedure is over and before the patient is awakened from anesthesia; blood sample will be taken, SpHb, PI and vital measurements (SpO2, Heart rate, NIBP, body temperature) will be recorded.
  Interventions: Device: Masimo Model RDS7A

INTERVENTIONS:
Device: Masimo Model RDS7A — Masimo monitoring platform equipped with Radical-7 Pulse CO-Oximeter fingertip probe for measurement non-invazive hemoglobin level (SpHb) an perfusion index (PI)

SUMMARY:
Pulse CO-Oximetry (Masimo Corp, Irvine, CA, USA) is a method that allows non-invasive continuous hemoglobin (Hb) measurement. This technology measures continuous Hb with a multi-wavelength spectrophotometric fingertip sensor.

Aim of investigators in this study is to make continuous Hb measurement with Pulse CO-Oximetry method in living liver donors, to compare these measurements with the laboratory results routinely taken during the operation, to determine the level of correlation for this patient group.

DETAILED DESCRIPTION:
Continuous Hb measurement with Pulse CO-Oximetry (SpHb) can be usefull for living liver donor and improve the quality of intraoperative care. This technology measures continuous Hb with a multi-wavelength spectrophotometric fingertip sensor.

The perfusion index (PI) is the ratio of the pulsatile blood flow to the nonpulsatile or static blood in peripheral tissue. Perfusion Index thus represents a noninvasive measure of peripheral perfusion that can be continuously and noninvasively obtained from a pulse oximeter. Changes in PI can also occur as a result of local vasoconstriction (decrease in PI) or vasodilatation (increase in PI) in the skin at the monitoring site. These changes occur with changes in the volumeof oxygenated bloodflow in the skin microvasculature. PI values can change due to surgical process and may affect SpHb measurement.

Aim of investigators in this study is to make continuous Hb measurement with Pulse CO-Oximetry method in living liver donors before and after surgery incision, to compare these measurements with the laboratory results routinely taken during the operation, to determine the level of correlation for this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing hepatectomy with general anesthesia

Exclusion Criteria:

* Patient's lack of consent, essential data missing, patient participating in other research projects, drug allergy, anesthetic complication story, excessive surgical bleeding, presence of disease that impairs peripheral circulation, use of vasoactive agents.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: According to ASA physical status classification system ASA 1-2 cases scheduled for hepatectomy for liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
CHb | Up to 14 weeks
  Correlation between non-invazive Hb measurement (measured by the masimo monitoring platform) and laboratuar Hb level.

SECONDARY OUTCOMES:
CPIS | Up to 14 weeks
  Correlation between Perfusion index (measured by the masimo monitoring platform) and surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu Univercity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No